CLINICAL TRIAL: NCT02555553
Title: Noom Monitor for Binge Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Noom Inc. (Industry); Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-1335
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Binge Eating Disorder
Keywords: Cognitive behavioral therapy guided self-help; Mobile Mental Health; Binge Eating; Cognitive Behavioral Therapy; Eating Disorder Treatment; Self-monitoring; Eating Disorders; Ecological Momentary Intervention
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): The control group for the RCT will be a "usual care" condition in which participants are free to seek any assistance for their ED during the study period.
- CBT-GSH with Noom Monitor (Experimental): Participation will include 12 weeks of guided cognitive-behavioral therapy- guided self help (CBT-GSH) with an MA-level health coach or nutritionist from the KPNW health plan. Patients will use a self-help book, Overcoming Binge Eating (2013) by Christopher Fairburn. The first session will last 60 minutes, and each subsequent session lasts 20-25 minutes. The first four sessions are weekly, with the subsequent four twice monthly. Self-monitoring will be conducted through Noom Monitor and individuals will receive a specialized set of instructions on how to use the monitor. Therapists will also be asked to check feedback report on clients before each session.
  Interventions: Behavioral: CBT-GSH with Noom Monitor

INTERVENTIONS:
Behavioral: CBT-GSH with Noom Monitor — This intervention is cognitive behavioral treatment with a smartphone application
  Arms: CBT-GSH with Noom Monitor

SUMMARY:
The purpose of the proposed Phase II STTR study is to test the primary efficacy of a novel mobile app, 'Noom Monitor,' in a large population of binge eaters in the Kaiser Permanente health care system relative to a well-established treatment as usual (TAU) control condition. Noom Monitor facilitates the delivery of CBT-GSH by utilizing a patient interface that increases adherence and provides between-session reminders of CBT-GSH principles. In addition, the Noom Monitor includes a therapist interface with weekly feedback to the provider about patient progress. This application has several primary objectives, including: (1) testing the real-world effectiveness of the Noom Monitor in a clinical setting, and (2) establishing a database of training materials for Noom Monitor. The knowledge gained from the current study will contribute to our understanding of the role of new emerging mobile technologies in augmenting existing treatments.

DETAILED DESCRIPTION:
Binge eating is a core maladaptive behavior characteristic of several forms of eating pathology, including bulimia nervosa (BN) and binge eating disorder (BED). These chronic conditions affect approximately 5% of the population, and cause significant psychosocial and physical impairment. However, a number of barriers prevent the implementation of effective treatments, including poor treatment adherence, a paucity of specialized therapists, and high rates of drop out. The guided self-help version of cognitive-behavior therapy (CBT-GSH) is a brief 8-session highly scalable treatment to reduce binge eating. Moreover, CBT-GSH is a cost-effective empirically supported treatment that has been demonstrated to reduce total health care costs.

Although CBT-GSH for BN and BED is effective, few individuals receive these treatments and the majority of other available treatments do not meet adequate standards for care for eating disorders. There are a number of reasons for why this is the case, but an important concern about CBT-GSH is participant burden. The primary CBT-GSH intervention is self-monitoring, a uniquely effective technique for reducing binge eating episodes; however, traditional self-monitoring is time-intensive and cumbersome because of its paper-and-pencil format. In addition, other behavioral strategies utilized in CBT-GSH (e.g., the development of regular eating) require a high degree of participant engagement outside of session. Novel technologies, such as those available with smartphones, offer potentially important means for reducing participant burden in the delivery of CBT-GSH. The purpose of the proposed is to test the primary efficacy of a novel mobile app, 'Noom Monitor' in a large population of binge eaters relative to a well-established treatment as usual (TAU) control condition. The investigative team developed these products via phase I study (R41-MH096435) to facilitate delivery of a cognitive-behavior therapy version of Guided Self-Help.

The efficacy and product development aims of this proposal will be used to support the commercial launch of Noom Monitor, a smartphone platform.

ELIGIBILITY:
Inclusion Criteria:

* Meets for DSM-5 BN or BED criteria
* Between the ages of 18 and 55
* Males and females
* BMI greater than 18.5 and less than 40
* Medical clearance in the case of reported purging or extreme exercise
* Free of psychiatric medication for at least 2 weeks prior to study or on a stable dose of medication for 4 weeks
* 1 year continuous enrollment in Kaiser Permanente Northwest health plan

Exclusion Criteria:

* Has undergone bariatric surgery
* Demonstrates need for higher level of care (e.g., very low weight (<18.5))
* Current comorbid substance dependence, bipolar or psychotic illness
* Current suicidal ideation
* Previously received Enhance Cognitive behavioral therapy or Cognitive behavioral therapy-guided self help
* Previously read Overcoming Binge Eating by Christopher Fairburn
* Purging and/or laxative use more than 2x a day on average over the last month.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Objective Binge Days | At 0 week
  Objective Binge Days - Objective binge days item of Eating Disorder Examination Scale version 16 (EDE-Q V6) - Frequency of days with objective binge episodes
Objective Binge Days | At 4 weeks
  Objective Binge Days - Objective binge days item of EDE-Q V6 - Frequency of days with objective binge episodes
Objective Binge Days | At 8 weeks
  Objective Binge Days - Objective binge days item of EDE-Q V6 - Frequency of days with objective binge episodes
Objective Binge Days | At 12 weeks
  Objective Binge Days - Objective binge days item of EDE-Q V6 - Frequency of days with objective binge episodes
Objective Binge Days | At 26 weeks
  Objective Binge Days - Objective binge days item of EDE-Q V6 - Frequency of days with objective binge episodes
Objective Binge Days | At 52 weeks
  Objective Binge Days - Objective binge days item of EDE-Q V6 - Frequency of days with objective binge episodes
Sum of Compensatory Episodes | At 0 week
  Sum of days where vomiting, laxative, or compulsive exercise occurs - sum of 3 items on EDE-Q v6
Sum of Compensatory Episodes | At 4 weeks
  Sum of days where vomiting, laxative, or compulsive exercise occurs - sum of 3 items on EDE-Q v6
Sum of Compensatory Episodes | At 8 weeks
  Sum of days where vomiting, laxative, or compulsive exercise occurs - sum of 3 items on EDE-Q v6
Sum of Compensatory Episodes | At 12 weeks
  Sum of days where vomiting, laxative, or compulsive exercise occurs - sum of 3 items on EDE-Q v6
Sum of Compensatory Episodes | At 26 weeks
  Sum of days where vomiting, laxative, or compulsive exercise occurs - sum of 3 items on EDE-Q v6
Sum of Compensatory Episodes | At 52 weeks
  Sum of days where vomiting, laxative, or compulsive exercise occurs -sum of 3 items on EDE-Q v6

SECONDARY OUTCOMES:
Clinical Impairment Assessment | At 0 week
  Full scale from 0-48, with higher score indicating more impairment
Clinical Impairment Assessment | At 4 weeks
  Full scale from 0-48, with higher score indicating more impairment
Clinical Impairment Assessment | At 8 weeks
  Full scale from 0-48, with higher score indicating more impairment
Clinical Impairment Assessment | At 12 weeks
  Full scale from 0-48, with higher score indicating more impairment
Clinical Impairment Assessment | At 26 weeks
  Full scale from 0-48, with higher score indicating more impairment
Clinical Impairment Assessment | At 52 weeks
  Full scale from 0-48, with higher score indicating more impairment
Personal Health Questionnaire | At 0 weeks
  Full scale from 0-24, with higher score indicating more depression
Personal Health Questionnaire | At 4 weeks
  Full scale from 0-24, with higher score indicating more depression
Personal Health Questionnaire | At 8 weeks
  Full scale from 0-24, with higher score indicating more depression
Personal Health Questionnaire | At 12 weeks
  Full scale from 0-24, with higher score indicating more depression
Personal Health Questionnaire | At 26 weeks
  Full scale from 0-24, with higher score indicating more depression
Personal Health Questionnaire | At 52 weeks
  Full scale from 0-24, with higher score indicating more depression
Quality of Life Scale | At 0 week
  Full scale from 16-112, with higher score indicating better health outcomes
Quality of Life Scale | At 4 weeks
  Full scale from 16-112, with higher score indicating better health outcomes
Quality of Life Scale | At 8 weeks
  Full scale from 16-112, with higher score indicating better health outcomes
Quality of Life Scale | At 12 weeks
  Full scale from 16-112, with higher score indicating better health outcomes
Quality of Life Scale | At 26 weeks
  Full scale from 16-112, with higher score indicating better health outcomes
Quality of Life Scale | At 52 weeks
  Full scale from 16-112, with higher score indicating better health outcomes
Eating Concern Subscale | At 0 week
  Eating concern subscale of the EDE-QV6 from 0-6 with higher score indicating worse health outcomes
Eating Concern Subscale | At 4 weeks
  Eating concern subscale of the EDE-QV6 from 0-6 with higher score indicating worse health outcomes
Eating Concern Subscale | At 8 weeks
  Eating concern subscale of the EDE-Q v6 from 0-6 with higher score indicating worse health outcomes
Eating Concern Subscale | At 12 weeks
  Eating concern subscale of the EDE-Q v6 from 0-6 with higher score indicating worse health outcomes
Eating Concern Subscale | At 26 weeks
  Eating concern subscale of the EDE-Q v6 from 0-6 with higher score indicating worse health outcomes
Eating Concern Subscale | At 52 weeks
  Eating concern subscale of the EDE-Q v6 from 0-6 with higher score indicating worse health outcomes
Dietary Restraint Subscale | At 0 week
  Dietary Restraint Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Dietary Restraint Subscale | At 4 weeks
  Dietary Restraint Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Dietary Restraint Subscale | At 8 weeks
  Dietary Restraint Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Dietary Restraint Subscale | At 12 weeks
  Dietary Restraint Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Dietary Restraint Subscale | At 26 weeks
  Dietary Restraint Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Dietary Restraint Subscale | At 52 weeks
  Dietary Restraint Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Shape Concern Subscale | At 0 week
  Shape Concern Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Shape Concern Subscale | At 4 weeks
  Shape Concern Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Shape Concern Subscale | At 8 weeks
  Shape Concern Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Shape Concern Subscale | At 12 weeks
  Shape Concern Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Shape Concern Subscale | At 26 weeks
  Shape Concern Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Shape Concern Subscale | At 52 weeks
  Shape Concern Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Weight Concern Subscale | At 0 Week
  Weight Concern Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Weight Concern Subscale | At 4 Weeks
  Weight Concern Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Weight Concern Subscale | At 8 Weeks
  Weight Concern Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Weight Concern Subscale | At 12 Weeks
  Weight Concern Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Weight Concern Subscale | At 26 Weeks
  Weight Concern Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Weight Concern Subscale | At 52 Weeks
  Weight Concern Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Global Eating Disorder Subscale | At 0 week
  Global Eating Disorder Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Global Eating Disorder Subscale | At 4 weeks
  Global Eating Disorder Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Global Eating Disorder Subscale | At 8 weeks
  Global Eating Disorder Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Global Eating Disorder Subscale | At 12 weeks
  Global Eating Disorder Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Global Eating Disorder Subscale | At 26 weeks
  Global Eating Disorder Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes
Global Eating Disorder Subscale | At 52 weeks
  Global Eating Disorder Subscale of the EDE-Q v6 from 0-6, with higher score indicating worse health outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hildebrandt, PsyD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Lynn DeBar, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

REFERENCES:
- [Derived] Hildebrandt T, Michaeledes A, Mayhew M, Greif R, Sysko R, Toro-Ramos T, DeBar L. Randomized Controlled Trial Comparing Health Coach-Delivered Smartphone-Guided Self-Help With Standard Care for Adults With Binge Eating. Am J Psychiatry. 2020 Feb 1;177(2):134-142. doi: 10.1176/appi.ajp.2019.19020184. PMID 32008396